CLINICAL TRIAL: NCT05821439
Title: The Effect of Menstruation on Food Preference and Balance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, hazal genc, Principal Investigator, Istanbul Medipol University Hospital
Other Study IDs: menstruation
Record Dates: First submitted 2023-04-06; First posted 2023-04-20 (Actual); Last update posted 2023-04-25 (Actual); Status verified 2023-04

CONDITIONS: Menstrual Cycle

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Premenstrual period: For the premenstrual period evaluation, the participants' 10 days before menstruation will be taken as a reference.
- Menstrual period: For the evaluation of the menstrual period, the first 3 days when symptoms are seen more will be taken as a reference.

SUMMARY:
Menstruation period, which is accepted as the symbol of fertility, and some problems related to this process covers half of a woman's life. During this period, various changes occur in the female body, especially in the endocrine system. These changes in the menstrual cycle can affect women physiologically and psychologically.

DETAILED DESCRIPTION:
Premenstrual syndrome (PMS) is an important health problem and negatively affects the quality of life of many women around the world. It usually begins 2 years after menarche and is known to worsen with age.It is known that approximately 80%-95% of women experience various degrees of PMS-related complaints. It has been reported that Premenstrual Syndrome can occur with more than 300 symptoms. The symptoms of PMS can be experienced in varying degrees, such as mild, moderate, and severe. The rate of those experiencing severe symptoms in PMS varies between 3-8%. Among the symptoms, psychological symptoms take the most important place. These; symptoms such as irritability, depression, anxiety, restlessness, nervousness, irritability, outbursts of anger and crying spells, feeling of loss of control, difficulty concentrating, laziness, insomnia or hypersomnia. The most common physical symptoms are joint, muscle, headache and abdominal pain, acne, edema, dizziness, libido and appetite changes, gastrointestinal disturbances, bloating, weight gain, breast fullness and tenderness.

ELIGIBILITY:
Inclusion Criteria

* Having completed the age of 18,
* Not over 45 years old and not in menopause,
* Not having any diagnosed psychological disease,
* It was determined as women who are healthy and have menstruation every month. Exclusion Criteria
* Individuals who menstruate with medical treatment every month,
* Individuals with lower extremity disability,

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Menstrual Period
Study Population: The study will be conducted using qualitative data with a total of 60 women in the 18-45 age group living in Turkey within 3 months following the ethics committee approval.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-04-23 (Actual); Primary Completion 2023-05-24 (Estimated); Study Completion 2023-07-21 (Estimated)

PRIMARY OUTCOMES:
star excursion balance test | one month
  On the previously prepared platform; There are 8 linear lines that form a star shape, arranged at an angle of 45 degrees between them. Before the test was administered to the individuals, necessary explanations were made and they were informed about the test. The individual to be tested was positioned to coincide with the very center of this shape. The untested leg was used to maintain the stability of the body in full contact with the ground. The tested leg, on the other hand, was asked to extend maximum in different directions and return to the starting position.
Food Record | one month
  Food records were evaluated in the "Nutrition Determine" program, and each participant received) amounts were calculated. Selections and intakes of nutrients will be evaluated. The Three-Factor Eating Questionnaire-Revised 18 Items (TFEQ-R18) consists of 18 items ona 4-point Likert scale (1 = definitely true, 2 = mostly true, 3 = mostly false, 4 = definitely false).Responses to each of the 18 items are summated into scale scores for cognitive restraint, uncontrolledeating, and emotional eating .igher scores in the respective scales areindicative of greater cognitive restraint, uncontrolled, or emotional eating.
General Anxiety Disorder | one month
  It is a test that evaluates the anxiety disorder of individuals with a short and self-reported way. It questions the emotions and mood changes experienced by individuals in the last 2 weeks. Each question of this test, which consists of 7 questions, has a 4-point Likert option. According to the scores obtained from the scale; 5,10,15 are used as cutoff points for mild, moderate and severe anxiety, respectively. In individuals with a total score of 10 and above, their anxiety should be investigated and confirmed by other methods. Score 0-4: Minimal Anxiety. Score 5-9: Mild Anxiety. Score 10-14: Moderate Anxiety. Score greater than 15: Severe Anxiety.
One Leg Standing Test | one month
  Before starting the test, the desired position was shown to the individuals and it will be explained in which cases the test will be invalid. This test was planned to be performed on both the right and left legs of the individuals. The desired position is for the untested leg; hip and leg flexed to 90 degrees, arms free, and the tested leg in full extension.
Premenstrual Syndrome Scale | one month
  Before answering the questions, individuals will be asked to think about the 7 days before menstruation. The scale consists of 44 questions in five-point Likert type.The lowest score is 44, and 220 is the highest. If the score (> 132)it will considered a positive Premenstrual Syndrome and as the score gets higher then indicate greater severity of symptoms during Premenstrual Syndrome .

SECONDARY OUTCOMES:
Three Factor Nutrition Questionnaire | one month
  With this questionnaire, which is used to evaluate the nutritional habits of individuals, our study measures the degree of conscious restriction of eating, the level of uncontrolled eating, and the degree of emotional eating.
Physical Activity Questionnaire | one month
  Physical activity level will be evaluated with the International Physical Activity .Scoring a HIGH level of physical activity on the IPAQ means your physical activity levels equate to approximately one hour of activity per day or more at least a moderate intensity activity level. intensity activities achieving a minimum total physical activity of at least 3000 MET minutes a week. Questionnaire (UFAA). The short form contains a total of 7 questions. Questionnaire; It allows us to obtain information about the time spent walking, during moderate and vigorous activities, and sitting. The measurement of all activities performed is based on the fact that each activity is performed for at least 10 minutes at a time. According to the total physical activity score, the physical activity levels of the participants are defined as "low, medium and high".

CONTACTS AND LOCATIONS:
Locations (1):
- HAZAL genç, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Souza LB, Martins KA, Cordeiro MM, Rodrigues YS, Rafacho BPM, Bomfim RA. Do Food Intake and Food Cravings Change during the Menstrual Cycle of Young Women? Rev Bras Ginecol Obstet. 2018 Nov;40(11):686-692. doi: 10.1055/s-0038-1675831. Epub 2018 Nov 28. PMID 30485899